CLINICAL TRIAL: NCT02990507
Title: Evaluation of an Advanced Virtual Exercise Environment Device (AVEED) for Use by Persons With Physical Disabilities
Brief Title: Advanced Virtual Exercise Environment Device for Use by Persons With Physical Disabilities
Acronym: AVEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laurie A Malone, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 123UAB
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Physically Disabled
Keywords: mobility impairment; virtual environment; exercise; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AVEED (Experimental): AVEED is composed of arm and leg cranks that can be used independently or together with a virtual exercise environment (VEE). Participants rotate arm and/or leg cranks under 4 conditions for 5 min each with a 5 min rest between: 1) Arm rotation with VEE, while sitting or standing (AVEED: Arm rotation, video display); 2) Arm rotation without VEE, while sitting or standing (AVEED: Arm rotation, without video display); 3) Leg rotation with arm-energy input to assist the legs with VEE, while sitting (AVEED: Leg rotation, arm-energy input, video display); 4) Leg rotation with arm-energy input to assist the legs without VEE, while sitting (AVEED: Leg rotation, arm-energy input, without video display). VEE controlled with voice commands, leaning, or keyboard buttons.
  Interventions: Other: AVEED: Arm rotation, video display; Other: AVEED: Arm rotation, without video display; Other: AVEED: Leg rotation, arm-energy input, video display; Other: AVEED: Leg rotation, arm-energy input, without video display

INTERVENTIONS:
Other: AVEED: Arm rotation, video display — Participants rotate arm cranks for 5 minutes then rest for 5 minutes.
Other: AVEED: Arm rotation, without video display — Participants rotate arm cranks for 5 minutes then rest for 5 minutes.
Other: AVEED: Leg rotation, arm-energy input, video display — Participants rotate leg cranks for 5 minutes then rest for 5 minutes.
Other: AVEED: Leg rotation, arm-energy input, without video display — Participants rotate leg cranks for 5 minutes then rest for 5 minutes.

SUMMARY:
An Advanced Virtual Exercise Environment Device (AVEED) has been developed that incorporates arm and leg ergometers in conjunction with a virtual reality interface. The purpose of this study is to examine participant perspectives regarding the virtual interface and exercise device combination with regard to usability, comfort, safety, rating of perceived exertion, and enjoyment.

DETAILED DESCRIPTION:
Individuals with physical disabilities show much lower rates of exercise participation than their able-bodied peers (Boslaugh et al. 2006, Preventing Chronic Disease). Much of the reason for the low rates of activity among this population come from the presence of barriers. Lack of motivation, lack of transportation, lack of accessible facilities and equipment, and cost are all factors that discourage exercise participation among those with disabilities (Rimmer et al. 2008, JRRD; Barfield and Malone 2013, JRRD). Based on these factors, there is a need for accessible enjoyable exercise options for people with physical disabilities. The AVEED is comprised of an ergometer with foot and hand pedals, and a visual display in front of the user that can show a variety of scenic pathways.

The AVEED builds on previous work that demonstrates the potential benefit of interactive exercise for those with physical disabilities. The present study will establish the potential of this device to provide an engaging moderate intensity exercise opportunity for persons with disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Mobility impairment, able to push a manual wheelchair

Exclusion Criteria:

* Individuals without a disability
* Individuals with vision loss that prevents them from seeing video elements on the screen
* Individuals with unstable cardiovascular conditions
* Individuals unable to push a manual wheelchair
* Individuals unable to understand study directions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Participant feedback | 2 days (approximately 48 hours) after enrolling
  Likert-style questions regarding ease of use, comfort, safety, and enjoyment related to using the device. Other questions will ask participants to compare the device with virtual interface to the device without the interface, as well as the likelihood of using their using the device if they had access to one.

SECONDARY OUTCOMES:
Exercise intensity | 2 days (approximately 48 hours) after enrolling
  Percent heart rate reserve (%HRR) is a measure of exercise intensity and is calculated as (HR - HRrest)/(HRmax - HRrest). Maximum HR can be estimated using the Karvonen formula which states HRmax = 220 - age. The participant's HR will be monitored in real time via a Bluetooth enabled device strapped to the chest. The goal is for the participant to input energy into the AVEED system and maintain a rate that produces a HRR of approximately 60%. Exercising at a rate of 60% of their age-predicted HRR, would establish them within the range of intensity for cardiovascular improvement. Verbal cues will be provided to ensure participants stay between 50-70% of HRR. If the participant is unable to sustain this intensity they will be allowed to rest for 1-2 minutes and then start again. Data recorded by the system will include continuous HR and energy output (watts).
Body orientation | 2 days (approximately 48 hours) after enrolling
  Video recordings will be used to assess how the participant's body is oriented in relation to the ergometer and their ease of use in rotating the cranks under the different conditions. the video will be scored using a 3 point likert scale: 1 being very poor body orientation to 3 being excellent orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Padalabalanarayanan, MS, Study Director — University of Alabama at Birmingham
Locations (1):
- Univerisity of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No